CLINICAL TRIAL: NCT06796192
Title: Assessment of the Protective Effect of Three Sunscreens on Visible Light Induced Pigmentation Compared with an Untreated Control Zone
Brief Title: Evaluate the Photoprotection Efficacy of Sunscreen Formulas Under Visible Light Exposure
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: EV1705-0432
Record Dates: First submitted 2025-01-14; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Study the Protection Potency of Sunscreen Products Against Pigmentation Induced by Visible Light Exposure on Healthy Back Skin
Keywords: Photoprotection; Sunscreen; Visible Light (VL); Pigmentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Product 1: The test product 1 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 2: The test product 2 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Product 3: The test product 3 was applied (2 mg/cm²) on the attributed zone according to the randomization list. The application was done during 4 consecutive days (From Day 1 to Day 4).
  Interventions: Other: Visible Light Exposure - Treated zones
- Untreated zone: non-treated control zone
  Interventions: Other: Visible Light Exposure - Untreated zone

INTERVENTIONS:
Other: Visible Light Exposure - Treated zones — The treated zones were exposed to Visible Light to induce skin pigmentation (144J/cm2), 15 minutes after application.
  Groups: Product 1; Product 2; Product 3
Other: Visible Light Exposure - Untreated zone — The untreated zone was exposed to Visible Light to induce skin pigmentation (144J/cm2), as the same time as the treated zones.
  Groups: Untreated zone

SUMMARY:
To evaluate the protective effect of three sunscreens on the pigmentation caused by visible light in comparison to an untreated control zone in healthy volunteers.

DETAILED DESCRIPTION:
The sunscreens usually used as photoprotectors are known to protect in the UV domain (UVB and UVA). However, until recently visible light (400-700 nm) was considered as devoid of any photobiological effects on cutaneous tissue. Over the last two decades, with the development of photodynamic therapies and various dermatological treatments using visible laser light, several studies have reconsidered the cutaneous effect of visible light on the skin, in particular the induction of pigmentation.

The aim of this study was to assess the ability of sunscreens with a protective efficacy in the UV domain to prevent the pigmentation induced by Visible Light.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject of both sexes, aged from 18 to 50 years, of phototype IIIb, IV or V on the Fitzpatrick scale (1988),
* Subject in good health having normal results for the physical examination and a medical antecedents compatible with the study requirements,
* Female subject of childbearing potential using a reliable means of contraception (contraceptive pill, contraceptive implant, IUD, bilateral tubal ligature/section, condoms) and accepting to not change her contraceptive status from at least one month prior to the start of the study and throughout the entire duration of the study,
* Female subject of non-childbearing potential, that was post-menopause (one year without menstruation), hysterectomy or bilateral ovariectomy,
* Subject having signed and dated the informed consent form before any study related action was initiated,
* Subject who was willing to follow the study procedures and to complete the study course,
* Subject affiliated to or beneficiary to a social security scheme (according to French legislation: Law 2004-806 and its implementing decree n°2006-477 of 26 April 2006).

Exclusion Criteria:

* Female who was pregnant or breastfeeding or who planned to become pregnant during the study,
* Subjects with an underlying pathology, or with a surgical, physical or medical status which, according to the investigator, could have interfered with the interpretation of the study results such as:

  1. Dermatological antecedents (e.g. acne, psoriasis, eczema, urticaria, etc.) or suspicion/antecedents of allergies to cosmetics,
  2. All systemic or local pathologies,
  3. Skin anomalies (scars, excessive hair, tattooing, etc.) on the test zones (back, middle section).
* Subjects having been excessively exposed to ultraviolet radiation (UV) natural (sun) or artificial (tanning salon) 2 months before the initial visit or who plans such an exposure during the study,
* Subjects having antecedents or currently presenting pathologies induced or aggravated by exposure to light or abnormal reactions to sunlight (e.g. : photosensitive dermatitis, polymorphous light reaction, benign summer light reaction, solar urticaria, systemic lupus erythematosus,dermatomyositis …),.
* Subjects having taken a systemic treatment for more than 5 days during the month preceding inclusion (steroids, non-steroidal anti-inflammatories such as aspirin, insulin, antihistamines, antihypertensives, antibiotics such as quinolones, tetracyclines, thiazides and fluoroquinolones, and all other photosensitising treatments) or all other treatments capable of inducing an abnormal response to UV or visible light (vitamin A derivatives, psoralen, aminolevulinic acid derivatives…) or planning to take these treatments during the study,
* Subjects having applied a local treatment on the back for more than 2 days during the 2 weeks preceding inclusion (steroids, non-steroidal anti-inflammatories, antihistamines, antibiotics) and all other cosmetic products in the previous 24 hours,
* Subject having antecedents of clinically significant allergy, particularly to study product components,
* Subjects requiring enhanced protection (deprived of liberty, minors, under guardianship),
* Subject being in a situation which, according to the Investigator, could interfere with an optimal participation in the study,
* Subject currently participating or having participated in another clinical trial during the month preceding inclusion,
* Subject unable to communicate efficiently with the Investigator or being unable to follow the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female volunteers from 18 to 50 years old with phototype III to V according to the Fitzpatrick scale
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Biophysical non-invasive assessment of skin color by using Chromameter® between the exposed zone (ZE) and non-exposed zone (ZNE) | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4, Day 5 (24 hours after each Visible Light exposure) and at Day 12..
  Individual Typologic Angle (ITA° - calculated value), • Pigmentation (Delta E, Delta L* and Delta b* - calculated values), • Erythema (Delta a* - calculated value).

SECONDARY OUTCOMES:
Clinical investigator's assessment by using clinical scale | At Day 1 before treatment (baseline), then Day 2, Day 3, Day 4, Day 5 (24 hours after each Visible Light exposure) and at Day 12..
  Visual scoring of pigmentation, using a pigmentation 11-point scale with 0 (No pigmentation), 1 (Doubtful), 2 (Very pale brown -), 3 (Very pale brown), 4 (Very pale brown +), 5 (Pale brown -), 6 (Pale brown), 7 (Pale brown +), 8 (Brown -), 9 (Brown), 10 (Brown +) Visual scoring of erythema, using an erythema 4-point scale with 0 (Absent), 0.5 (Doubtful), 1 (Weak but well-defined erythema), 2 (Moderate), 3 (Severe)
Safety / Local Tolerance | From the informed consent signature date until the end of the study (Day 12)
  Safety was assessed by recording Adverse Events, including cutaneous reactions (local intolerance) assessed using the following 5-point score system:
  0 (no sign/symptom of local intolerance); 0.5 (doubtful sign/symptom of local intolerance); 1 (mild sign/symptom of local intolerance); 2 (moderate sign/symptom of local intolerance); 3 (severe sign/symptom of local intolerance)

CONTACTS AND LOCATIONS:
Locations (1):
- CPCAD (Centre de Pharmacologie Clinique Appliquée à la Dermatologie), Nice, France

IPD SHARING:
Plan to Share IPD: No